CLINICAL TRIAL: NCT01904344
Title: NXT_SLEEP: the Development of a Next Generation Sleep Monitoring Platform
Brief Title: Clinical Validation of New Breathing Sensors in Patients With Respiratory Insufficiency
Acronym: NXT_SLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: iMinds (Industry)
Responsible Party: Principal Investigator, Wilfried De Backer, MD PhD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PML_NXT_SLEEP
Record Dates: First submitted 2013-07-08; First posted 2013-07-22 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Respiratory Patients
Keywords: Sleep; Sleep- related breathing disorders; Respiratory pathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sensor testing and validation (Other)
  Interventions: Device: Sensor testing and validation

INTERVENTIONS:
Device: Sensor testing and validation

SUMMARY:
The NXT_SLEEP study, bringing together industry partners, research groups and (home) care providers, tackles will develop a next generation sleep-monitoring platform that consists of less obtrusive sensors, and that delivers complete and useful information regarding the physiological parameters relevant for sleep-related breathing disorders.

These new and innovative sensors need to be validated in a clinical setting where they will be benchmarked with the classical sleep monitoring systems. In order to compare the novel sensors with the classical monitoring system, the investigators use existing technologies that capture simultaneously the acquired signals of different physiological parameters relevant for sleep-related breathing disorders.

DETAILED DESCRIPTION:
Sleep-related breathing disorders are recognized as major risk factors for mortality due to their effect on the cardiovascular system. Currently, these sleeping disorders are diagnosed using polysomnography (PSG), which is a sleep test that monitors different physiological signals such as heart rate, respiration, ECG, muscle tone and eye movement.

Although polysomnography is an important diagnostic tool for sleep medicine, it is an uncomfortable and costly procedure, especially when multiple nights of observation are required. In order to reduce costs and improve patients comfort, different home monitoring systems (using different numbers and type of sensors) have been introduced to the market, but those focus especially on self-screening and collect general sleep information. In addition to increasing comfort and reducing costs, the diagnostic capabilities of PSG need to be enhanced. This can be achieved by adding novel sensors that may capture new information and improve the measurement of vital physiological parameters during sleep

ELIGIBILITY:
Inclusion Criteria:

* Patients who are hospitalized for their respiratory disease
* Written informed consent obtained

Exclusion Criteria:

* Patients with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially comprise the results of interpretation of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in breathing pattern during sleep by a movement sensor | During 5 nights
  New innovative sensors will measure breathing pattern during the night, simultaneously with the classical monitoring systems in order to validate the new sensors.

SECONDARY OUTCOMES:
Change in ECG | During 5 nights
Change in end tidal carbon dioxide fraction | During 5 nights

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium